CLINICAL TRIAL: NCT06049693
Title: Iron Prehabilitation and Perioperative Infectious Diseases of Endometrial Cancer Patients
Brief Title: Iron Prehabilitation in Endometrial Cancer
Acronym: IROGYN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Nikolaos Thomakos, Associate Professor of Obstetrics and Gynecology, National and Kapodistrian University of Athens
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 129/20
Record Dates: First submitted 2023-04-25; First posted 2023-09-22 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Endometrial Cancer; Perioperative Complication; Prehabilitation
MeSH Terms: conditions — Endometrial Neoplasms | interventions — ferrous gluconate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iron supplementation (Experimental): Iron supplementation will be provided in the form of ferrous gluconate 300mg twice a day for a period of 1 month
  Interventions: Drug: Ferrous Gluconate 300 MG
- Control (No Intervention): Control patients will be recruited on the ground of no form of iron prehabilitation

INTERVENTIONS:
Drug: Ferrous Gluconate 300 MG — Ferrous Gluconate 300 MG twice a day
  Arms: Iron supplementation

SUMMARY:
Endometrial cancer patients often have iron deficiency anemia before surgery, which can be effectively treated with oral iron supplementation. Anemia and blood transfusions have been previously associated with perioperative infectious diseases. In the present study the investigators will evaluate the impact of perioperative iron supplementation on the incidence of perioperative infections.

DETAILED DESCRIPTION:
Prehabilitation has a multimodal conception based on three fundamental pillars: improvement of the patient's physical condition, nutritional optimization and other measures such as smoking cessation and correction of anemia.

As in the case of multimodal rehabilitation protocols, the actions of prehabilitation programs have synergistic effects, that is, small changes that, by themselves, do not have clinical significance but when added up, they produce a significant improvement in the postoperative evolution of patients.

Surgical site infections (SSIs) are considered to be the most common nosocomial infections among surgical patients and constitute a heavy and potentially preventable economic burden on health care providers. Although the impact of blood transfusion on the risk of SSI remains controversial, several studies have shown that anemia and transfusion predispose to postoperative bacterial infections.

In the present study the investigators seek to evaluate the impact of per os iron prehabilitation on perioperative outcomes of endometrial cancer patients, including need for transfusion and infectious morbidity.

ELIGIBILITY:
Inclusion Criteria:

Women with endometrial cancer enrolled in the surgical list

Exclusion Criteria:

Women with endometrial cancer requiring immediate surgery due to life-threatening hemorrhage

Ages: 18 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with endometrial cancer will be recruited
Enrollment: 156 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with surgical site infection | Postoperatively (up to 30 days)
  Participants will be followed-up to determine the incidence of postoperative surgical site infection
Required blood transfusions per participant and aggregated mean differences | Perioperatively (up to 10 days)
  The number of perioperative (intraoperative and postoperative) blood transfusions per patient will be monitored and compared among the two groups.

SECONDARY OUTCOMES:
Number of participants with other postoperative infections | Postoperatively (up to 30 days)
  Participants will be followed-up to determine the incidence of other postoperative infectious morbidity (other than surgical site infection)
Duration of hospitalization per participant | Postoperatively (until patient exit) up to 30 days
  The duration of hospitalization per participant will be monitored.
Onset of adjuvant treatment per participant | Postoperatively up to 24 weeks
  The interval between surgery and adjuvant treatment will be monitored.
Survival rates of included participants | Postoperatively (at 3 years postoperatively)
  Patients will be screened for recurrence of disease and their survival status will be screened at 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- First department of Obstetrics and Gynecology, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared upon reasonable request

REFERENCES:
- [Background] Amstad G, Geiger J, Werlen L, Montavon C, Heinzelmann V. Perioperative management with ferric carboxymaltose and tranexamic acid to reduce transfusion rate in gynaecological carcinoma surgery (TRANAFER-Study): study protocol for a single-blind, monocentre, randomised trial. BMJ Open. 2022 Sep 26;12(9):e057381. doi: 10.1136/bmjopen-2021-057381. PMID 36167367
- [Background] Tyan P, Taher A, Carey E, Amdur R, Messersmith C, Robinson HN, Gu A, Vargas MV, Moawad GN. Effect of Perioperative Transfusion on Postoperative Morbidity Following Minimally Invasive Hysterectomy for Benign Indications. J Minim Invasive Gynecol. 2020 Jan;27(1):200-205. doi: 10.1016/j.jmig.2019.03.021. Epub 2019 Mar 28. PMID 30930213
- [Background] Fung PLP, Lau VNM, Ng FF, Leung WW, Mak TWC, Lee A. Perioperative changes in haemoglobin and ferritin concentrations from preoperative intravenous iron isomaltoside for iron deficiency anaemia in patients with colorectal cancer: A pilot randomised controlled trial. PLoS One. 2022 Jun 30;17(6):e0270640. doi: 10.1371/journal.pone.0270640. eCollection 2022. PMID 35771891
- [Background] Bath M, Viveiros A, Schaefer B, Klein S, Pammer LM, Wagner S, Lorenz A, Rugg C, Gasser E, Ninkovic M, Panzer M, Pertler E, Fries D, Tilg H, Weiss G, Petzer V, Ofner-Velano D, Zoller H. Impact of preoperative anemia, iron-deficiency and inflammation on survival after colorectal surgery-A retrospective cohort study. PLoS One. 2022 Jul 27;17(7):e0269309. doi: 10.1371/journal.pone.0269309. eCollection 2022. PMID 35895618